CLINICAL TRIAL: NCT05125549
Title: Fasting, Comparative, Open-label, Randomized, Four-period, Two-sequence, Bioequivalence Study of Сlopidogrel Bisulfate Film-coated Tablets, 75 mg (JSC Farmak, Ukraine) vs Plavix® 75 mg Film-coated Tablets in Healthy Adult Subjects
Brief Title: Fasted Bioequivalence Study of Clopidogrel Film-coated Tablets, 75 mg in 48 Healthy, Adult Male and Female Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joint Stock Company "Farmak" (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FK-CLP
Record Dates: First submitted 2021-11-16; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics
Keywords: bioequivalence; pharmacokinetics; generic drugs; Clopidogrel; Film-coated Tablets
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Сlopidogrel bisulfate film-coated tablets, 75 mg (JSC Farmak, Ukraine)
  Interventions: Drug: Сlopidogrel bisulfate film-coated tablets, 75 mg (JSC Farmak, Ukraine)
- Treatment B (Active Comparator): Plavix® 75 mg film-coated tablets (Sanofi Winthrop Industrie, France)
  Interventions: Drug: Plavix® 75 mg film-coated tablets (Sanofi Winthrop Industrie, France)

INTERVENTIONS:
Drug: Сlopidogrel bisulfate film-coated tablets, 75 mg (JSC Farmak, Ukraine) — One film-coated tablet was administrated orally with 240 ml of water after an overnight fast
  Other Names: Trombonet
  Arms: Treatment A
Drug: Plavix® 75 mg film-coated tablets (Sanofi Winthrop Industrie, France) — One film-coated tablet was administrated orally with 240 ml of water after an overnight fast
  Arms: Treatment B

SUMMARY:
This study was designed to compare bioequivalence of the Test Product Clopidogrel bisulfate, film-coated tablets, 75 mg (JSC Farmak, Ukraine) and Reference Product Plavix® 75 mg film-coated tablets (Sanofi Winthrop Industrie, France) in healthy male and female volunteers under fasting conditions.

DETAILED DESCRIPTION:
An open, comparative, randomized, four-period, two- sequence, two-way crossover clinical trial to evaluate the Bioequivalence of Single Doses of Test Product Clopidogrel bisulfate, film-coated tablets, 75 mg (JSC Farmak, Ukraine) and Reference Product Plavix® 75 mg film-coated tablets (Sanofi Winthrop Industrie, France) in healthy adult male and female volunteers under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and non-pregnant and no breast-feeding females1), ≥18 and ≤50 years of age (on the day of Informed Consent). Caucasian race.
* Subject had provided his/her written informed consent before the start of any screening procedures.
* Subject was available for the whole study and to follow all the requirements of the study protocol.
* Body Mass Index (BMI) 18.5 to 30.0 kg/m2, inclusive (on the day of screening).
* Subject without any acute or chronic diseases of the cardiovascular system, neuroendocrine system, kidney, liver, gastrointestinal tract, respiratory system.
* Subjects in good health, as determined by screening medical history, physical examination, vital signs assessments (pulse rate, systolic and diastolic blood pressure, and body temperature) and 12-lead electrocardiogram (ECG). Minor deviations outside the reference ranges were acceptable, if deemed not clinically significant by the Investigator
* The results of fluorography are within normal ranges (no more than 10 months before inclusion in the study).
* Sitting blood pressure is within normal ranges: 100 -140 mm Hg for systolic PB, 55 -95 mm Hg. for diastolic blood pressure (BP) at screening;
* Acceptance of use of contraceptive measures during the whole study by both female and male subjects.
* Non-smoker
* Subject is available to comply with the general dietary restrictions throughout the study.

Exclusion Criteria:

* History of severe allergy or allergic reactions to the study Investigational Medicinal Product (IMP), its excipients or related drugs.
* Aggravated allergic history
* History of any clinically significant disease or disorder or surgical intervention which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* A positive result of Hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), and / or (human immunodeficiency virus) HIV or syphilis tests during screening procedure.
* A positive results of urine drug of abuse test (amphetamine, methamphetamine, morphine, marijuana, cocaine).
* Positive result of alcohol breath test
* Positive urine cotinine test
* The values of the standard parameters of the laboratory and instrumental examinations are outside the normal range and are clinically relevant or require additional examination and interpretation.
* Pregnancy (positive urine pregnancy test result in women)
* Lactation period (for women).
* Acute infectious diseases in less than 28 days before the first dosing.
* Use of any medication for a period of 14 days before the first dosing.
* Donation of blood within 30 days before the first dosing.
* Participation in any other clinical study during last 90 days.
* Other reasons when participation of a volunteer in the study is undesirable in the opinion of the Investigator.

Ages: 18 Years to 50 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Сmax | up to 36 hours post-administration
  maximum plasma concentration observed
AUC0-t | up to 36 hours post-administration
  area under the plasma concentration versus time curve calculated by the trapezoidal rule from sampling time zero to sampling time of the last measurable plasma concentration

SECONDARY OUTCOMES:
tmax | up to 36 hours post-administration
  the time of the maximum plasma drug concentration

OTHER OUTCOMES:
λz | up to 36 hours post-administration
  apparent first-order elimination
t1/2 | up to 36 hours post-administration
  the elimination or terminal half-life
AUC0-∞ | up to 36 hours post-administration
  area under the plasma concentration versus time curve from time zero to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Udovytskyi, Study Chair — Joint Stock Company "Farmak"
Locations (1):
- Clinical and Diagnostics Center of National University of Pharmacy (NUPh)., Kharkiv, Ukraine

IPD SHARING:
Plan to Share IPD: No